CLINICAL TRIAL: NCT07352696
Title: Effects of Combined High-Intensity Aerobic Training and Resistance Training on Cardiovascular and Metabolic Health in Psoriatic Arthritis
Brief Title: Combined High-Intensity Aerobic Training and Resistance Training in Psoriatic Arthritis
Acronym: PsA-HIIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vastra Gotaland record 286312
Record Dates: First submitted 2025-12-15; First posted 2026-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Treatment versus care as usual
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Cardiorespiratory and strength training, 2-3 sessions per week for a total of 12 weeks.
  Interventions: Behavioral: Exercise program
- Control group (No Intervention): Care as usual, plus individualized counseling for health-promoting physical activity

INTERVENTIONS:
Behavioral: Exercise program — The exercise program includes two supervised sessions per week combining high-intensity interval training and strength training, plus one additional non-supervised aerobic session. The target of the high intensity intervals is 90%-95% of heart rate maximum. The strength training of major muscle groups includes 2-3 sets of 8-10 repetitions.
  Arms: Exercise group

SUMMARY:
The goal of this randomised controlled trial is to evaluate the effects of a 12-week intervention comprising high-intensity interval aerobic training and strength training on cardiovascular function, metabolic health profile and inflammation in patients with Psoriatic arthritis. A secondary goal is to assess the intervention´s impact on physical fitness, pain, fatigue, and health-related quality of life, and to explore long-term maintenance of exercise following completion of the intervention. We hypothesize that 12 weeks of combined high-intensity interval aerobic training and strength training will improve cardiometabolic health, inflammation, and enhance physical fitness, fatigue, pain and quality of life in Psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Psoriatic arthritis disease according to the CASPAR (Classification Criteria for Psoriatic Arthritis) criteria
* Age range 18-65 years
* Stable medication on anti- rheumatic drugs for >3 months prior to inclusion and throughout the first 3 months of the study

Exclusion Criteria:

* Cardiovascular disease
* Severe hypertension
* Diabetes type I
* Chronic obstructive pulmonary disease or other severe pulmonary diseases
* Arthroplasty of large joints, lower extremities
* Severe functional impairment precluding participation in high-intensity aerobic exercise
* Inability to perform a cardiopulmonary exercise testing (CPET)
* Pregnancy
* BMI ≥35 kg/m²
* Ongoing or planned initiation (within 3 months) of structured weight reduction therapy, pharmacological obesity treatment, or bariatric bypass surgery
* Already participating in regular exercise at high intensity (BORG ≥15) for >1 hour/ week during the past 6 months
* Inability to understand and read Swedish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary function | Baseline and 3 month
  Change in maximum oxygen uptake (VO2ml/min/kg). Higher value indicate better cardiorespiratory capacity.
Cardiopulmonary function | Baseline and 9 month
  Change in maximum oxygen uptake (VO2ml/min/kg). Higher value indicate better cardiorespiratory capacity)

SECONDARY OUTCOMES:
Waist circumference | Baseline and 3 months
  Change in waist circumference (cm) measured with a tape measure midway between the lower rib and iliac crest. A waist measurement of 80 centimeters or more for women and 94 centimeters or more for men indicate increased risk for diseases related to overweight.
Waist circumference | Baseline and 9 months
  Change in waist circumference (cm) measured with a tape measure midway between the lower rib and iliac crest. A waist measurement of 80 centimeters or more for women and 94 centimeters or more for men indicate increased risk for diseases related to overweight.
Body mass index (BMI) | Baseline and 3 months
  Change in Body Mass Index (BMI). Weight and height will be combined to report BMI (kg/m2). A higher score indicate higher relative weight.
Body mass index (BMI) | Baseline and 9 months
  Change in Body Mass Index (BMI). Weight and height will be combined to report BMI (kg/m2). A higher score indicate higher relative weight.
Body composition | Baseline and 3 months
  Change in total leanmass (%) and fatmass (%) assessed with Bioelectrical Impedance Analysis. Higher value indicate higher total leanmass and fatmass
Body composition | Baseline and 9 months
  Change in total leanmass (%) and fatmass (%) assessed with Bioelectrical Impedance Analysis. Higher value indicate higher total leanmass and fatmass
Triglycerides | Baseline and 3 months
  Change in triglycerides (mmol/L)
Triglycerides | Baseline and 9 months
  Change in triglycerides (mmol/L)
High-density lipoprotein cholesterol (HDL-C) | Baseline and 3 months
  Change in high-density lipoprotein cholesterol (HDL-C) (mmol/L)
High-density lipoprotein cholesterol (HDL-C) | Baseline and 9 months
  Change in high-density lipoprotein cholesterol (HDL-C) (mmol/L)
Low-density lipoprotein cholesterol (LDL-C) | Baseline and 3 months
  Change in low-density lipoprotein cholesterol (LDL-C) (mmol/L)
Low-density lipoprotein cholesterol (LDL-C) | Baseline and 9 months
  Change in low-density lipoprotein cholesterol (LDL-C) (mmol/L)
Total cholesterol | Baseline and 3 months
  Change in total cholesterol (mmol/L)
Total cholesterol | Baseline and 9 months
  Change in total cholesterol (mmol/L)
Glycosylation level of hemoglobin (HbA1c) | Baseline and 3 months
  Glycosylation level of hemoglobin (HbA1c) (mmol/mol)
Glycosylation level of hemoglobin (HbA1c) | Baseline and 9 months
  Glycosylation level of hemoglobin (HbA1c) (mmol/mol)
Homeostatic model assessment of insulin resistance (HOMA IR) | Baseline and 3 monhts
  Measure of insulin resistance (fasting glucose (mmol/L) and fasting insulin (mIU/ L) will be combined to report Homeostatic model assessment of insulin resistance (HOMA IR).
Homeostatic model assessment of insulin resistance (HOMA IR) | Baseline and 9 months
  Measure of insulin resistance (fasting glucose (mmol/L) and fasting insulin (mIU/ L) will be combined to report Homeostatic model assessment of insulin resistance (HOMA IR).
Erythrocyte Sedimentation Rate (ESR) | Baseline and 3 months
  Change in level of erytrocyte rate (ESR) (mm/h). Higher score indicate higher degree of inflammation.
Erythrocyte Sedimentation Rate (ESR) | Baseline and 9 months
  Change in level of erytrocyte rate (ESR) (mm/h). Higher score indicate higher degree of inflammation.
C-Reactive Protein (CRP) | Baseline and 3 months
  Change in level of of high sensitivity CRP (mg/L). Higher score indicate higher inflammation.
C-Reactive Protein (CRP) | Baseline and 9 months
  Change in level of of high sensitivity CRP (mg/L). Higher score indicate higher inflammation.
Cytokine levels | Baseline and 3 months
  Change in inflammatory cytokines such as Interleukin-6 (pg/mL), interleukin-10 (pg/mL), tumour necrosis factor-alpha (pg/mL).
Disease activity | Baseline and 3 months
  Change in Disease Activity index for PSoriatic Arthritis (DAPSA) score. Calculated by summing 66/68 joints (swollen, tender), patient global assessment (VAS), pain (VAS)and CRP). A higher value indicates a higher disease activity. (Minimum: 0=no disease activity, >28= high disease activity).
Disease activity | Baseline and 9 months
  Change in Disease Activity index for PSoriatic Arthritis (DAPSA) score. Calculated by summing 66/68 joints (swollen, tender), patient global assessment (VAS), pain (VAS)and CRP). A higher value indicates a higher disease activity. (Minimum: 0=no disease activity, >28= high disease activity).
Muscle function lower extremities | Baseline and 3 months
  Change in the one minute sit-to-stand test (STS). Higher numbers of complete rises indicate better muscle function in lower extremities.
Muscle function lower extremities | Baseline and 9 months
  Change in the one minute sit-to-stand test (STS). Higher numbers of complete rises indicate better muscle function in lower extremities.
Handgrip strength | Baseline and 3 months
  Change in grip strength measured with a dynamometer (newton). Higher value indicate better grip strength.
Handgrip strength | Baseline and 9 months
  Change in grip strength measured with a dynamometer (newton). Higher value indicate better grip strength.
Activity limitations | Baseline and 3 months
  Change in Health Assessment Questionnaire (HAQ) (0-3). A higher score indicates more activity limitations
Activity limitations | Baseline and 9 months
  Change in Health Assessment Questionnaire (HAQ) (0-3). A higher score indicates more activity limitations.
Physical function | Baseline and 3 months
  Change in the Bath Ankylosing Spondylitis Functional Index (BASFI) (0-10). Higher score indicate more physical limitations
Physical function | Baseline and 9 months
  Change in the Bath Ankylosing Spondylitis Functional Index (BASFI) (0-10). Higher score indicate more physical limitations
Physical activity | Baseline and 3 months
  Change in self-reported weekly physical activity assessed with the International Physical Activity Questionnaire (IPAQ)-Short Form. Time spent in low, moderate, and vigorous activity is summed within each intensity category. (According to WHO guidelines, ≥150 minutes of moderate or ≥75 minutes of vigorous activity per week qualifies as health-enhancing physical activity).
Physical activity | Baseline and 9 months
  Change in self-reported weekly physical activity assessed with the International Physical Activity Questionnaire (IPAQ)-Short Form. Time spent in low, moderate, and vigorous activity is summed within each intensity category. (According to WHO guidelines, ≥150 minutes of moderate or ≥75 minutes of vigorous activity per week qualifies as health-enhancing physical activity).
Attitude to exercise | Baseline and 3 months
  Change in exercise believe assessed with the Exercise Health Beliefs questionnaire (20-100), Higher score represents stronger exercise beliefs.
Attitude to exercise | Baseline and 9 months
  Change in exercise believe assessed with the Exercise Health Beliefs questionnaire (20-100), Higher score represents stronger exercise beliefs.
Emotional experience of exercise | Baseline and 3 months
  Change in the Physical Activity Enjoyment Scale (PACES) (18-126). Higher score indicate higher degreee of enjoyment and pleasure related to exercising.
Emotional experience of exercise | Baseline and 9 months
  Change in the Physical Activity Enjoyment Scale (PACES) (18-126). Higher score indicate higher degreee of enjoyment and pleasure related to exercising.
Sleep quality | Baseline and 3 months
  Change in Pittsburgh Sleep Quality Index (PSQI) (0-21), Higher score indicate worse sleep quality.
Sleep quality | Baseline and 9 months
  Change in Pittsburgh Sleep Quality Index (PSQI) (0-21), Higher score indicate worse sleep quality.
Fatigue | Baseline and 3 months
  Change in The Multiple Fatigue Inventory (MFI-20), 4-20 for each subscale, Higher score indicates a higher degree of fatigue.
Fatigue | Baseline and 9 months
  Change in The Multiple Fatigue Inventory (MFI-20), 4-20 for each subscale, Higher score indicates a higher degree of fatigue
Pain intensity | Baseline and 3 months
  Visual Analogue Scale (VAS) (0-100), Higher score indicate worse pain.
Pain intensity | Baseline and 9 months
  Visual Analogue Scale (VAS) (0-100), Higher score indicate worse pain.
Global health | Baseline and 3 months
  Change in Visual Analogue Scale (VAS) (0-100), Higher score indicate worse health
Global health | Baseline and 9 months
  Change in Visual Analogue Scale (VAS) (0-100), Higher score indicate worse health
Health related quality of life | Baseline and 3 months
  Change in the 36-item Short Form Health Survey (SF-36) questionnare (0-100). A higher score indicate better health related quality of life
Health related quality of life | Baseline and 9 months
  Change in the 36-item Short Form Health Survey (SF-36) questionnare (0-100). A higher score indicate better health related quality of life
The impact of the disease on quality of life | Baseline and 3 months
  Change in the Dermatology Life Quality Index (DLQI) (0-30). Higher score indicate worse impairment
The impact of the disease on quality of life | Baseline and 9 months
  Change in the Dermatology Life Quality Index (DLQI) (0-30). Higher score indicate worse impairment
Mental health | Baseline and 3 months
  Change in the Hospital and Anxiety Depression Scale (HADS) for anxiety and depression (0-21). A higher score refers to a higher degree of distress.
Mental health | Baseline and 9 months
  Change in the Hospital and Anxiety Depression Scale (HADS) for anxiety and depression (0-21). A higher score refers to a higher degree of distress.
Disease related symptoms | Baseline and 3 months
  Patient Global Impression of Change (PGIC) scale (0-7) to adress changes in symtoms. Rating from very much improved (7) to very much worse (1).
Disease related symptoms | Baseline and 9 months
  Patient Global Impression of Change (PGIC) scale (0-7) to adress changes in symtoms. Rating from very much improved (7) to very much worse (1).
Enthesites | Baseline and 3 months
  Change in the Entesiter MASES entesit index. Palpation of 13 body sites for tenderness. (0= no tenderness, 1= tenderness presented) Higher scores indicate more widespread/tender enthesitis.
Enthesites | Baseline and 9 months
  Change in the Entesiter MASES entesit index. Palpation of 13 body sites for tenderness. (0= no tenderness, 1= tenderness presented). Higher scores indicate more widespread/tender enthesitis.
Skin involvement | Baseline and 3 months
  Skin involvement evaluated using the Body surface area (BSA), percentage of total body surface affected by lesions.
Skin involvement | Baseline and 9 months
  Skin involvement evaluated using the Body surface area (BSA), percentage of total body surface affected by lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Annelie Bilberg, Assoc. Prof., Principal Investigator — Sahlgrenska University hospital, Gothenburg
Locations (2):
- Sweden (2):
  - Sahlgrenska University hospital, Gothenburg
  - Skaraborgs sjukvård, Skövde, Skövde

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in a publication are available from the principal investigator (P.I.) on reasonable request. Access will be determined based on reasonable request and in accordance with the ethical approval
Time Frame: The data will become available as following, starting 6 months after publication and end 5 years after publication.
Access Criteria: The requests will be reviewed by the P.I. and the steering committee. Study plans on meta-analyses generating new knowledge on exercise in persons with rheumatic diseases will be approved.